CLINICAL TRIAL: NCT01475396
Title: Clinical Study on the Effect of Physical Activity on Cognition and Memory in the Elderly
Brief Title: The Effect of Physical Activity on the Brain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Exercise_Neuromod
Record Dates: First submitted 2011-11-07; First posted 2011-11-21 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Aerobic Exercise; Anaerobic Exercise; Unchanged Condition
Keywords: exercise; physical activity; cognition; brain; aging; BDNF
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: exercise
- Anaerobic Exercise (Experimental)
  Interventions: Behavioral: exercise
- Unchanged condition (No Intervention)

INTERVENTIONS:
Behavioral: exercise
  Arms: Aerobic Exercise; Anaerobic Exercise

SUMMARY:
Physical activity is thought to increase overall body functions and to decrease cardiovascular and stroke risk factors. Now the question arose, wether enhanced exercise could also exert positive influence on cognition in the aging brain. Therefore, 50 to 80 years old healthy subjects take part in a prospective study with regular sports activity during 6 months. Cognitive functions are detected with sensitive neuropsychological outcome measures, further investigations include MRT of the head, lactat- and other physical measures as well as detailed serum profiles. As a hypothesis, enhanced physical activity is suggested to predict better cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years old
* healthy
* lesser activity

Exclusion Criteria:

* regular physical activity
* diabetes
* stroke
* heavy smoking, drinking,
* BMI < 20
* MMSE < 25

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-03; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change of reaction times in ms in a motor learning task after 6 months of intervention/control condition | 6 months
Change of delayed memory scores in #of words in a Verbal learning task after 6 months of intervention/control condition | 6 months
Change of performance in ms in a reaction time task after 6 months of intervention/control condition | 6 months
Change of relative regional grey matter volumes in % measured by T1-weighted MRI after 6 months of intervention/control condition | 6 months

SECONDARY OUTCOMES:
Change of physical measurements (ECG)/fitness assessments (lactate) after 6 months of intervention/control condition | 6 months
Change of BDNF blood serum levels in ng/dl after 6 months of intervention/control condition | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flooel, MD, Principal Investigator — University Hospital of Muenster; Stefan Knecht, MD, Study Director — University Hospital of Muenster
Locations (1):
- University Hospital of Muenster, Münster, North Rhine-Westphalia, Germany